CLINICAL TRIAL: NCT05859360
Title: Functional Exercise Training With Adolescents and Young Adults With Cerebral Palsy: Follow Up Study
Brief Title: Functional Exercise Training in Cerebral Palsy: Follow Up
Acronym: FITCP
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Alice Minghetti, Dr. sc. med., University of Basel
Other Study IDs: FITCP: Follow Up
Record Dates: First submitted 2023-05-04; First posted 2023-05-16 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: functional training; strength; cardiovascular health; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Functional Performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Trained CP: Adolescents and young adults with CP who have continued their regular training after completing the pilot study.
  Interventions: Other: Physical performance and cardiovascular health measures
- Untrained CP: Adolescents and young adults with CP who have not continued their regular training after completing the pilot study.
  Interventions: Other: Physical performance and cardiovascular health measures
- Trained Peers: Healthy peers who perform high-intensity strength training on a regular basis.
  Interventions: Other: Physical performance and cardiovascular health measures
- Untrained Peers: Healthy peers who do not perform high-intensity strength training on a regular basis.
  Interventions: Other: Physical performance and cardiovascular health measures

INTERVENTIONS:
Other: Physical performance and cardiovascular health measures — * Retinal vessel analysis
  * Muscle ultrasound
  * Knee extension
  * Voluntary activation
  * spiroergometry

SUMMARY:
The goal of this cross-sectional study is to compare able-bodied peers to adolescents and young adults with cerebral palsy (CP) who have been regularly performing high-intensity functional training for almost two years.

The main research question is: is structured, long-term exercise training able to compensate strength and cardiovascular deficits in adolescents with CP compared to able-bodied peers?

DETAILED DESCRIPTION:
The pilot study investigating the effects of a functional exercise training in adolescents and young adults with cerebral palsy (CP) showed increases in strength, power, daily function as well as cardiovascular health. In order to establish the origin of the improvements and its broader effects, we wish to conduct follow-up measurements to the pilot study. These follow-up measurements would establish whether the positive changes in physical performance are due to neural or muscular changes (or both), and shed more light on how therapy should be performed and prescribed in adolescents with CP. Additionally, we wish to measure their aerobic capacity as well as examine their microvascular health. For this cross-sectional analysis, the participants of the CP-FIT Pilot Study who continued to train on a regular basis will be compared to age-matched peers in order to establish whether their strength and fitness deficits compared to peers can be compensated through structured and progressive functional exercise training.

ELIGIBILITY:
Inclusion Criteria:

CP Individuals:

* Diagnosis of CP.
* Between 14 and 26 years of age.
* Gross Motor Functional Classification System (GMFCS): I-II.
* Cognitive abilities must include: Ability to verbally or non-verbally communicate pain or discomfort; Ability to attend testing and; ability to understand and follow instructions. All included participants are capable of making decisions on their own and no not show any signs of mental or cognitive limitations.

Healthy peers:

- Between 14 and 26 years of age.

Exclusion Criteria:

CP Individuals:

* Any surgery or botulinum toxin treatment within 6 months prior to the measurements or scheduled during study period. Other medications can be continued as prescribed by the participants' physician.
* Known cardiovascular or pulmonary diseases that have not received medical clearance to participate in physical exercise.
* Uncontrolled seizures or epilepsy.
* Inability to conform to the above mentioned cognitive and physical abilities.

Healthy peers:

* Diagnosis of congenital heart defects, pulmonary diseases or any neuromuscular disorders or diseases.
* Diagnosis of any acute diseases.

Ages: 14 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The group adolescents with CP consists of individuals from the CP-FIT pilot study who have both continued or discontinued their training after study completion. Healthy peers are age- and sex-matched able-bodied peers.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Maximum knee extension force | 20 minutes
  Maximum force of knee extension in relation to body weight

SECONDARY OUTCOMES:
Microvascular health | 5 minutes
  Static retinal vessel analysis
Voluntary activation | 15 minutes
  Maximum force able to voluntarily activate
Spiroergometry | 20 minutes
  Cardiopulmonary test on bicycle ergometer
Muscle architecture | 10 minutes
  Ultrasound of defined muscle groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport, Exercise and Health, University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No
No IPD will be made public. Group data will be analysed for publication after study completion.